CLINICAL TRIAL: NCT00161850
Title: Follow-up Study to Investigate the Safety and Immunogenicity of a Third Vaccination With Three Different Antigen Concentrations of FSME IMMUN NEW in Children Aged 1 to 6 Years
Brief Title: FSME IMMUN NEW Follow-up to Study 199 in Children Aged 1 to 6 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 206
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Encephalitis, Tick-borne
MeSH Terms: conditions — Encephalitis, Tick-Borne | interventions — Vaccines

INTERVENTIONS:
Biological: Tick-Borne Encephalitis (TBE) Vaccine (Inactivated)

SUMMARY:
The purpose of this study is to investigate the safety and immunogenicity of the third vaccination with one of three different concentrations of a TBE vaccine in all subjects who completed two vaccinations in one of the three treatment groups of Baxter study 199 (a dose-finding study to investigate the safety and immunogenicity of two vaccinations with FSME IMMUN NEW in healthy subjects aged 1 to 6 years).

ELIGIBILITY:
Inclusion Criteria:

All volunteers who participated in Baxter study 199 and received two vaccinations will be invited to participate. Male and female children will be eligible for participation in this study if:

* They received two vaccinations with one of the three different dosages of FSME IMMUN NEW during the course of Baxter study 199
* Written informed consent from the legal guardian is available.

Exclusion Criteria:

There are no specific exclusion criteria for this study entry. However volunteers will be assessed for eligibility to receive a third vaccination.

Volunteers will be excluded from vaccination and consecutive visits in this study if they:

* Are not clinically healthy, (i. e. the physician would have reservations vaccinating with FSME IMMUN NEW outside the scope of a clinical trial)
* Have already been administered a third TBE vaccination elsewhere after the two vaccinations in Baxter study 199
* Have had an allergic reaction to one of the components of the vaccine since the last vaccination in Baxter study 199
* Suffer from a disease (e.g. autoimmune disease) or are undergoing a form of treatment (e.g. systemic corticosteroids, chemotherapeutics) that can be expected to influence immunological functions
* Have received banked human blood or immunoglobulins within one month of study entry
* Are known to be HIV positive (a special HIV test is not required for the purpose of the study) since the last visit of Baxter study 199
* Have had a vaccination against yellow fever and / or Japanese B-encephalitis since the last visit in Baxter study 199
* Had received an investigational new drug within 6 weeks prior to study start

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 615
Dates: Start 2002-02; Study Completion 2002-08

CONTACTS AND LOCATIONS:
Overall Officials: Baxter BioScience Investigator, Principal Investigator — Baxter Healthcare Corporation
Locations (25):
- Grieskirchner Strasse 17, Wels, Austria
- Germany (24):
  - Neuschwanstein Strasse 5, Augsburg
  - Marktplatz 33, Bad Saulgau
  - Hauptstrasse 9, Bietigheim-Bissingen
  - Salzgasse 11, Calw
  - Mohrenstrasse 8, Coburg
  - Bahnhofstrasse 1, Elzach
  - Rheinstrasse 1a, Ettenheim
  - Ehlerstrasse 17, Friedrichshafen
  - Peter-Seifert Strasse 5, Gersfeld
  - Solothumer Strasse 2, Heilbronn
  - Hauptstrasse 240, Kehl
  - Schwarzwald Strasse 20, Kirchzarten
  - Altoettinger Strasse 3, Landsberg
  - Rastatter Strasse 7, Mannheim-Secken
  - Wilhelmstrasse 25, Metzingen
  - Dohmbuehler Strasse 8, Nuremberg
  - Glogauer Strasse 15, Nuremberg
  - Tuchbergstrasse 2, Oberndorf/Neckar
  - Wilhelmstrasse 7, Offenburg
  - Asternweg 11a, Offenburg
  - Bergstrasse 27, Rottweil
  - Berneckstrasse 19, Schramberg
  - Hauptstrasse 11, Tegernsee
  - Broner Platz 6, Weingarten